CLINICAL TRIAL: NCT06470399
Title: AI-Guided (GenAIS TM) Versus Standard Physician-Guided Dietary Supplementation for Managing Metabolic Syndrome: A Randomized Controlled Study
Brief Title: AI-Guided (GenAIS TM) Versus Standard Physician-Guided Dietary Supplementation for Managing Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW017
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome
Keywords: AI-guided dietary supplementation; Metabolic parameters improvement; Genetic profiling; metabolic profiling
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Standard therapy group
- AI-Guided Group (Experimental)
  Interventions: Other: AI-Guided Group

INTERVENTIONS:
Other: Standard therapy group — Participants receive DS prescriptions from a physician based on current standard practices, which include biochemical markers, genetic data, and metabolic profiles.
  Arms: Control Group
Other: AI-Guided Group — Participants receive DS prescriptions determined by GenAIS, is an AI system that considers genetic data, metabolic profiles, biochemical markers, and patient history.
  Arms: AI-Guided Group

SUMMARY:
The study "AI-Guided (GenAIS TM) Versus Standard Physician-Guided Dietary Supplementation for Managing Metabolic Syndrome" aimed to compare the effectiveness of AI-guided dietary supplement (DS) prescriptions versus standard physician-guided prescriptions in managing metabolic syndrome. This 6-month randomized controlled trial included 160 participants diagnosed with metabolic syndrome. Participants were divided into two groups: one received DS based on physician judgment, and the other based on GenAIS AI system analysis. Primary outcomes focused on changes in metabolic parameters, while secondary outcomes included individual components of metabolic syndrome, inflammation levels, body weight, and adherence to the DS regimen. Data collection involved genetic, metabolic, and clinical profiling, with ethical considerations ensuring participant confidentiality and informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years.
* Diagnosed with metabolic syndrome, defined by the presence of at least three of the following criteria:
* Waist circumference > 102 cm (men) or > 88 cm (women).
* Triglycerides ≥ 150 mg/dL.
* HDL cholesterol < 40 mg/dL (men) or < 50 mg/dL (women).
* Blood pressure ≥ 130/85 mm Hg.
* Fasting glucose ≥ 100 mg/dL. • Willingness to provide genetic and metabolic data.

Exclusion Criteria:

* Significant renal, hepatic, or cardiovascular diseases.
* Use of dietary supplements that affect metabolic parameters within the last 3 months.
* Pregnancy or breastfeeding.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Composite Metabolic Syndrome Score | 6 months
  This includes measuring and tracking changes in the five main components of metabolic syndrome: waist circumference, triglycerides, high-density lipoproteins ( HDL) cholesterol, blood pressure, and fasting glucose. These components are central to the definition of metabolic syndrome and are commonly used to assess the efficacy of interventions. The Composite Metabolic Syndrome Score combines multiple metabolic risk factors and typically ranges from 0 (optimal) to 5 (worst), with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Waist Circumference change in cm | 6 months
Triglycerides change in mg/dl | 6 months
HDL Cholesterol change in mg/dl | 6 months
Blood Pressure change in mmHg | 6 months
Fasting Glucose in mg/dl | 6 months
High-Sensitivity C-Reactive Protein change | 6 months
Body Weight change in kg | 6 months
body mass index (BMI) change | 6 months
Incidence of any Adverse Effects | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia